CLINICAL TRIAL: NCT01518127
Title: Intravitreal Bone Marrow-Derived Stem Cells in Patients With Macular Degeneration
Acronym: AMDCELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rubens Camargo Siqueira, MD,PhD - Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sao Paulo University
Record Dates: First submitted 2011-09-20; First posted 2012-01-25 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Age Related Macular Degeneration and Stargartd
Keywords: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Intervention Model Description: intravitreal injection of autologous bone marrow stem cells
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell group (Experimental): intravitreal injection of autologous bone marrow stem cells
  Interventions: Other: intravitreal injection of autologous bone marrow stem cells

INTERVENTIONS:
Other: intravitreal injection of autologous bone marrow stem cells — intravitreal injection of autologous bone marrow stem cells
  Other Names: Cell Therapy

SUMMARY:
The purpose of this study is to evaluate the behavior of intravitreal injection of of autologous bone marrow stem cells in patients with age related macular degeneration.

DETAILED DESCRIPTION:
A prospective phase I/II, nonrandomized open-label study of agen related macular degeneration and Stargartd patients with best-corrected ETDRS visual acuity (BCVA) worse than 20/200. Standardized ophthalmic evaluation will be perform at baseline and at weeks 1, 4,12 and 24 (±1) following intravitreal injection of 10 x 106 bone marrow stem cells/ 0,1ml . Three measures will be used to evaluate the short-term safety of intravitreal of bone marrow stem cells: 1) severe visual loss, defined as a drop in 15 letters on ETDRS visual acuity scale; 2) decrease in ERG response; 3) decrease in 5 square degrees on visual field; secondary safety outcomes : 1) increase in intra-ocular inflammation defined herein as anterior chamber cells and flare higher than 3+ for more than 1 month after injection according to a classification described elsewhere ; 2) decrease in CMT more than 50um; 3)genesis of abnormal tissues (teratomas) or tumors; 4) qualitative changes in retinal or choroidal perfusion, like macular nonperfusion. Secondary outcome measures will be used to evaluate the short-term efficiency of intravitreal of Bone Marrow Stem Cells: 1) improvement in ERG response; 2) increase in visual field: 3) increase in CSMT > 50um and not related to macular edemar or choroidal neovascularization; 4) increase > 5 letters on BCVA

ELIGIBILITY:
Inclusion Criteria:

* Male or female AMD and Stargartd patients 18 to 80 years old, inclusive.
* In either eye, diagnosis of geographic atrophy or choroidal neovascularization due to AMD
* ETDRS best corrected visual acuity of 60 letters or worse in the study eye.

Exclusion Criteria:

* Retinal disease other than AMD in study eye which, in the investigator's opinion, may pose a safety risk or interfere with the study.
* Choroidal neovascularization due to a cause other than AMD.
* In the study eye, media opacity that interferes with fundus imaging or is likely to require surgery during the study period.
* Any of the following treatments to the study eye within 14 days prior to dosing: ranibizumab (Lucentis), bevacizumab (Avastin), pegaptanib (Macugen), or other VEGF inhibitor; OR likely requirement for one of the above treatments within 14 days of LFG316 administration.
* Any of the following within 30 days prior to dosing: photodynamic therapy treatment in the study eye; extrafoveal or juxtafoveal thermal laser photocoagulation in the study eye; systemic or topical (ophthalmic) steroid use in the study eye; bacterial keratitis in the study eye; OR intraocular surgery (including cataract surgery) in the fellow eye.
* Any of the following within 90 days prior to dosing: intraocular surgery (including cataract surgery) in the study eye; OR intravitreal or periocular corticosteroid injection in the study eye.
* Participation in another interventional clinical study, or use of any experimental treatment for AMD or any other investigational new drug within 12 weeks prior to the start of study treatment. Clinical trials solely involving over-the-counter vitamins, supplements, or diets will not exclude the patients from study participation.
* Any medical condition likely to interfere with the patient's participation in the study, or likely to cause serious adverse events during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
ETDRS Visual acuity change | Day 1 to Day 365
  Primary safety outcome included visual acuity loss of 15 or more ETDRS letters after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rubens C Siqueira, MD,PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Rubens Siqueira Research Center, São José do Rio Preto, São Paulo, Brazil